CLINICAL TRIAL: NCT04032847
Title: An Open-Label, Multi-Centre Phase I/IIa Study Evaluating the Safety and Clinical Activity of Neoantigen Reactive T Cells in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: ATL001 in Patients With Advanced Unresectable or Metastatic NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Achilles Therapeutics UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATX-NS-001
Record Dates: First submitted 2019-07-17; First posted 2019-07-25 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Following lymphodepletion with enhanced host conditioning, infusion of cell therapy product ATL001, followed by a low dose regimen of IL- 2.
  Interventions: Biological: ATL001
- Cohort B (Experimental): Following lymphodepletion with enhanced host conditioning, infusion of cell therapy product ATL001 in combination with a checkpoint inhibitor, followed by a low dose regimen of IL- 2.
  Interventions: Biological: ATL001; Drug: Pembrolizumab
- Cohort C (Experimental): Following lymphodepletion with enhanced host conditioning, infusion of cell therapy product ATL001, followed by a higher dose regimen of IL-2.
  Interventions: Biological: ATL001

INTERVENTIONS:
Biological: ATL001 — ATL001 infusion
Drug: Pembrolizumab — Checkpoint inhibitor
  Arms: Cohort B

SUMMARY:
This is a first-in-human, open-label, multi-centre, phase I/IIa study to characterise the safety and clinical activity autologous clonal neoantigen reactive T cells (cNeT) administered intravenously in adults with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a first-in-human, open-label, multi-centre, phase I/IIa study to characterise the safety and clinical activity of autologous clonal neoantigen reactive T cells (cNeT) administered intravenously in adults with advanced non-small cell lung cancer (NSCLC).

Patients will initially enter the study for procurement of tumour materials required to manufacture ATL001.

Following manufacture of ATL001, the product will be given back to eligible patients following lymphodepletion. Patients will continue to be followed up for a minimum of 5 years, as part of a separate Long Term Follow Up Protocol, or, if the separate protocol is not available at the study site, within this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at 18-75 years old.
2. Patients must have confirmed diagnosis of non-small cell lung cancer that is considered to be smoking related.
3. Patient is considered medically fit to undergo procurement of starting material and ATL001 administration procedures.
4. ECOG Performance Status 0-1.
5. Adequate organ function per the laboratory parameters defined in the protocol.
6. Anticipated life expectancy ≥ 6 months at the time of tissue procurement.
7. Measurable disease according to RECIST 1.1 criteria.

Additional Inclusion Criteria will apply as per the protocol.

Exclusion Criteria:

1. Patients with untreated, symptomatic or progressing CNS metastases. Lesions should be clinically and radiologically stable for 2 months after treatment and should not require steroids.
2. Patients with hepatitis B or C, human immunodeficiency virus infection (HIV1/2), syphilis or HTLVI/II infection.
3. Patients for whom there is documented evidence of an actionable tumour driver oncogene mutation (EGFR, ALK or ROS-1) at the time of initial screening. Patients who have progressed on standard targeted therapies, or for whom no approved targeted treatments are available, are not excluded.
4. Patients requiring immunosuppressive treatments.
5. Patients requiring regular steroids at dose higher than prednisolone 10mg/day (or equivalent)
6. Patients with superior vena cava syndrome.
7. Patients with clinically significant, progressive, and/or uncontrolled renal, hepatic, haematological, endocrine, pulmonary, cardiac, gastroenterological or neurological disease.
8. Patients with a history of immune mediated central nervous system toxicity, or a history of ≥ Grade 2 diarrhoea/colitis within the past 6 months caused by previous immunotherapy.
9. Patients with an active concurrent cancer or a history of cancer within the past 3 years (except for in situ carcinomas, early prostate cancer with normal Prostate- Specific Antigen (PSA) or non-melanomatous skin cancers)
10. Patients with a history of organ transplantation
11. Patients who have previously received any investigational cell or gene therapies

Additional Exclusion Criteria will apply as per the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Achilles Therapeutics
Locations (19):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France
- Germany (2):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Instituto de Investigación Sanitaria Fundación Jimenez Díaz, Madrid
  - Centro Integral Oncologico Clara Campal Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (9):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge
  - The Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds
  - University College London Hospitals (UCLH) NHS Foundation Trust, University College Hospital, London
  - Guys and St Thomas' NHS Foundation Trust, Guy's Hospital, London
  - The Christie NHS Foundation Trust, Christie Hospital, Manchester
  - Manchester University NHS Foundation Trust, Wythenshawe Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust, Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please be advised that Cohort B was not formally opened therefore, no patients were enrolled into this arm.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 22 (Refers to patients treated with ATL001 in Cohort A) | 0 | 5 (Refers to patients treated with ATL001 in Cohort C)
Completed | 0 | 0 | 0
Not Completed | 22 | 0 | 5
Not completed — Study termination by sponsor | 8 | 0 | 4
Not completed — Death | 12 | 0 | 0
Not completed — Progressive disease | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Cohort B never opened
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 22 | 0 | 5 | 27
Age, Customized [Count of Participants; unit: Participants]
  Age: <65 years | 19 |  | 1 | 20
  Age: >=65 years | 3 |  | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 |  | 1 | 11
  Male | 12 |  | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 1 |  | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 18 |  | 4 | 22
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 3 |  | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 1 | 4
  United Kingdom | 11 |  | 1 | 12
  France | 3 |  | 0 | 3
  Germany | 4 |  | 2 | 6
  Spain | 1 |  | 1 | 2
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: (kg/m^2)] | 26.75 (5.818) |  | 27.10 (4.256) | 26.81 (5.490)
Baseline ECOG performance status [Count of Participants; unit: Participants] — The ECOG (Eastern Cooperative Oncology Group) performance score is a widely used scale to assess a patient's level of functioning, particularly in cancer clinical trials.
  This assessment was performed at the Baseline Screening period by the clinical research teams when they reviewed their patients.
  Score 0: Fully active, able to carry out all pre-disease performance without restrictions.
  Score 1: Restricted in physically strenuous activity but ambulatory and able to perform light work.
  Participants
    Grade 0 | 8 |  | 2 | 10
    Grade 1 | 14 |  | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Treatment Emergent Adverse Events (TEAEs) to Evaluate Safety and Tolerability
Description: Evaluate TEAEs and serious AEs, by incidence, severity and relationship to ATL001
Time Frame: 62 months due to early termination
Population: Cohort B never opened.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 22 | 0 | 5
Participants
  TEAEs | 21 |  | 5
  TEAEs related to any component of study treatment | 19 |  | 5
  Lymphodepletion related TEAEs | 16 |  | 4
  ATL001 related TEAEs | 16 |  | 4
  IL-2 related TEAEs | 16 |  | 5
  Serious TEAEs | 6 |  | 0
  Serious TEAEs related to any component of study treatment | 2 |  | 0
  Serious Lymphodepletion related TEAEs | 1 |  | 0
  Serious ATL001 related TEAEs | 1 |  | 0
  Serious IL-2 related TEAEs | 0 |  | 0
  TEAEs with CTCAE grade >= 3 | 16 |  | 5
  TEAEs with CTCAE grade >= 3 related to any component of study treatment | 14 |  | 4
  Lymphodepletion related TEAEs with CTCAE grade >= 3 | 12 |  | 4
  ATL001 related TEAEs with CTCAE grade >= 3 | 4 |  | 2
  IL-2 related TEAEs with CTCAE grade >= 3 | 6 |  | 3
  TEAEs leading to death | 0 |  | 0
  SAEs | 8 | 0 | 0

2. Secondary Outcome: Disease Assessment for Change From Baseline in Tumour Size
Description: Evaluate the clinical activity of ATL001 in patients with advanced NSCLC using change from baseline in tumour size at week 6 , week 12 and best overall change from baseline, as assessed by investigator and independent central review (ICR)
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

3. Secondary Outcome: Disease Assessment for Time to Response (TTR) From ATL001 Infusion
Description: Evaluate the endpoint of TTR by the investigator and ICR, per RECIST v1.1 and im-RECIST
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

4. Secondary Outcome: Disease Assessment for Objective Response Rate (ORR)
Description: Evaluate the endpoint of overall response rate (ORR), as assessed by investigator and ICR, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and immune modified RECIST( im-RECIST).
  RECIST v1.1 (Response Evaluation Criteria in Solid Tumors) is a standardized system for measuring tumor response to treatment in clinical trials. Tumors are assessed by imaging (e.g., CT or MRI) based on changes in size. Responses are categorized as:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): ≥30% reduction in the sum of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD).
  Progressive Disease (PD): ≥20% increase in the sum of target lesions, or appearance of new lesions.
  These criteria help assess the efficacy of treatments in solid tumors supported by im-RECIST in immunotherapy.
Time Frame: Every 6 weeks for 6 months, then every 3 months (up to 62 months due to early termination)
Population: No patients treated in Cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 22 | 0 | 5
Participants
  Responders | 2 | 0 | 0
  Non-Responders | 20 | 0 | 5

5. Secondary Outcome: Disease Assessment for Duration of Response (DoR). The DoR is Defined as the Time From the Date of First Documented Response Until the Date of Documented Disease Progression or Death
Description: Evaluate the endpoint of DOR by the investigator and ICR, per RECIST v1.1 and im-RECIST
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

6. Secondary Outcome: Disease Assessment for Disease Control Rate (DCR)
Description: Evaluate the endpoints of DCR as assessed by the investigator and ICR per RECIST v1.1 and im-RECIST
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

7. Secondary Outcome: Disease Assessment for Progression-Free Survival (PFS)
Description: Evaluate the efficacy endpoints of PFS as assessed by the investigator and ICR per RECIST v1.1 and im-RECIST
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival (OS)
Description: Evaluate OS by the investigator
Time Frame: Every 6 weeks for 6 months, then every 3 months for a maximum of 84 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Each patient that received ATL001 would have been followed up for 24 months, to withdrawal of consent or death. Patients would then continue to be followed up for a minimum of 5 years as part of long term follow up. The study was terminated early due to sponsor decision. The Median follow-up period was 12 weeks (range: 3 - 48 weeks).
Arm/Group | Cohort A | Cohort C
All-Cause Mortality (participants affected / at risk) | 14/22 | 1/5
Serious Adverse Events (participants affected / at risk) | 8/22 | 0/5
Other Adverse Events (participants affected / at risk) | 22/22 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=22) | Cohort C (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=22) | Cohort C (N=5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (18) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 3 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (5) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 14 (18) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Fatigue (General disorders) | 11 (11) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (11) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 6 (7) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 2 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 10 (11) | 2 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (8) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 9 (11) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (12) | 2 (3)
Pyrexia (General disorders) | 13 (15) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 4 (6) | 1 (1)
Asthenia (General disorders) | 3 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 4 (5)
Oedema (General disorders) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (2)
Chills (General disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 4 (5)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Range of other disclosure agreements across study sites. Following multi-center publication of the Study results made by Sponsor, the Institution and/or Principal Investigator may publish data or results from the Study provided the Sponsor is given 45 to 90 days to review and/or make comments and suggestions where pertinent.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04032847/Prot_SAP_000.pdf